CLINICAL TRIAL: NCT00012623
Title: Improving Service Delivery Through Access Points
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: ACC 97-068
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension; Angina; Diabetes
MeSH Terms: conditions — Hypertension; Angina Pectoris; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
CBOCs represent one of VA's main managed care strategies for shifting the focus of care from the inpatient to the outpatient setting and for improving the health of our nation's veterans. Hypothesis-driven research is critically needed to test the basic assumptions motivating the expansion of CBOCs throughout the VA health care system.

DETAILED DESCRIPTION:
Background:

CBOCs represent one of VA's main managed care strategies for shifting the focus of care from the inpatient to the outpatient setting and for improving the health of our nation's veterans. Hypothesis-driven research is critically needed to test the basic assumptions motivating the expansion of CBOCs throughout the VA health care system.

Objectives:

The purpose was to determine how increased geographic access to primary care services affects service use and costs. Two specific aims addressed were: 1) to determine how CBOCs impact the service use of all existing users and existing users with the following ambulatory care sensitive conditions (ACSC): alcohol dependence, angina, chronic obstructive pulmonary disease (COPD), depression, diabetes and hypertension; and 2) to describe how CBOCs affect the workload and costs of the VA health care system from the VISN's perspective.

Methods:

A quasi-experimental pre-post study design with intervention and reference groups was employed to compare service use and costs in the 18 months following the establishment of a new CBOC. Fifteen CBOCs from 11 VISNs were included in the analysis. For specific aim 1, the intervention group was defined as existing users in the catchment area of a new CBOC and the reference group was defined as matched existing users outside CBOC catchment areas. Multivariate statistical regression analyses were used to estimate the impact of residing within the CBOC catchment area on use and cost in the post-period, controlling for patient casemix and use/cost in the 18 month pre-period. For specific aim 2, the intervention group was defined as zip codes in the catchment area of a new CBOC and the reference group was defined as matched zip codes outside CBOC catchment areas. Average use and costs for all users, existing users and new users from intervention zip codes and reference zip codes were compared.

Status:

Complete.

ELIGIBILITY:
Inclusion Criteria:

Subjects must live in the catchment area of a specified CBOC and have been diagnosed with a tracer condition.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39481 (Estimated)
Dates: Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Fortney, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Washington, United States

REFERENCES:
- [Result] Fortney JC, Maciejewski ML, Warren JJ, Burgess JF Jr. Does improving geographic access to VA primary care services impact patients' patterns of utilization and costs? Inquiry. 2005 Spring;42(1):29-42. doi: 10.5034/inquiryjrnl_42.1.29. PMID 16013585